CLINICAL TRIAL: NCT04582552
Title: A Real-world Study of Clinical Markers for PARP Inhibitors in Epithelial Ovarian Cancer
Brief Title: The Clinical Markers for PARP Inhibitors-related Efficacy in Ovarian Cancer
Acronym: ROMP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiaoxiang Chen (Other)
Responsible Party: Sponsor-Investigator, Xiaoxiang Chen, Academic secretary of gynecological oncology Committee of Jiangsu anti cancer association, Jiangsu Cancer Institute & Hospital
Organization: Jiangsu Cancer Institute & Hospital (Other)
Other Study IDs: JiangsuCH
Record Dates: First submitted 2020-10-05; First posted 2020-10-09 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Ovarian Cancer; Clinical Marker; PARP Inhibitor
Keywords: Ovarian caner, PARP inhibitor, Clinical marker
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Poly(ADP-ribose) Polymerase Inhibitors; olaparib; niraparib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ovarian cancer patients treated with PARP inhibitors: PARP inhibitors therapy until disease progression
  Interventions: Drug: PARP inhibitors

INTERVENTIONS:
Drug: PARP inhibitors — Ovarian cancer patients with PARP inhibitors according to the NCCN guideline and their instructions.
  Other Names: Lynparza, Zejula

SUMMARY:
Epithelial ovarian cancer (EOC) is the most lethal gynecological malignancy. PARP inhibitors(PARPi) are an important progress in EOC treatment. The available evidence suggests that BRCAmt or HRD-positive is an effective biological marker for PARPi. However, in our previous clinical observation, it was found that the tumor burden may be the potential clinical markers PARPi. We intend to develop a real-world study to confirm the potential clinical markers and explore new clinical markers for PARPi.

DETAILED DESCRIPTION:
This study intends to conduct a systematic real-world study to observe the relationship between the clinical characteristics of EOC patients and the efficacy of PARPi based on our existing research foundation and stratified analyse these correlations by BRCA and HRD status.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects join the study voluntarily and sign informed consent;
2. Female subjects are older than 18 years;
3. ECOG(Eastern Cooperative Oncology Group) physical status score is 0-2;
4. Life expectancy≥3 months;
5. Histologically confirmed FIGO(International Federation of Gynecology and Obstetrics ) III/IV ovarian cancer, fallopian tube cancer, or primary peritoneal cancer; Participants must have high-grade serous or endometrioid histology;
6. Patients should test for BRCA gene and will perform test for HRD status if who harbor BRCAwt in the same laboratory designated by the researcher;
7. Patients received PARP inhibitor as maintenance therapy or monotherapy for more than four weeks.

Exclusion Criteria:

1. Personnel involved in the formulation or implementation of the research plan;
2. Patient participated in other clinical trails using other experimental drugs at the same time as the study;
3. The subjects had other malignant diseases in past 2 years, except skin squamous cell carcinoma, basal-like carcinoma, breast intraductal carcinoma in situ, or cervical carcinoma in situ;
4. Previous or currently diagnosed myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML);
5. Patients who are pregnant or lactation, or who plan to become pregnant during study treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ovarian cancer patients treated with PARP inhibitor in the real word.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Through study completion, an average of 1 year
  ORR is defined as the proportion of participants achieving complete response (CR) or partial response (PR) as assessed by RECIST1.1.
Progression Free Survival (PFS) | Through study completion, an average of 1 year
  PFS is defined as the time in months from the date of first study drug administration to the date of first documentation of progressive disease (PD) or death as assessed by RECIST1.1.
Duration of Response (DOR) | Through study completion, an average of 1 year
  DOR is defined as the time from the first date of response until the date of first documented progression.
Disease Control Rate (DCR) | Through study completion, an average of 1 year
  DCR is defined as the proportion of participants achieving complete response (CR), partial response (PR) or stable disease (SD) according to RECIST1.1.
Adverse events (AEs) | Through study completion, an average of 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE 5.0 to further describe safety and assess toxicities encountered with the use of the proposed treatment regimen in participants.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxiang Chen, MD,PhD, Study Chair — Jiangsu Cancer Institute & Hospital; Jing Ni, MD, Principal Investigator — Jiangsu Cancer Institute & Hospital
Locations (1):
- Xiaoxiang Chen, MD,PhD, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Contact Prof. Chen and Dr. Ni for primary data.